CLINICAL TRIAL: NCT07174791
Title: Fully Versus Partially Guided All on Four Implants Placement Immediately Loaded by Maxillary and Mandibular Screw Retained Prosthesis: A Radiographic and Photogrammetric Measurement of Accuracy of Implant Position and Passivity of Superstructures
Brief Title: Fully Versus Partially Guided Implants Placement: Measurement of Accuracy of Implant Position and Passivity of Superstructures.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed shady, Assistant professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: A03010024RP
Record Dates: First submitted 2025-06-22; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Completely Edentulous; Implant Assesment
Keywords: Guided surgery; semi-guided surgery; full arch implants; photogrammetry
MeSH Terms: interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Intervention Model Description: According to the virtual 3D planning and surgical guide designing for implant instalment, patients will be randomly divided into two equal treatment groups (4 patients for each) as follows:
  Group (I): partially- guided (PG) implant instalment Group (II): fully- guided (FG)implant instalment both groups will be subjected to:
  1. cone beam computed tomography to evaluate peri-implant alveolar bone loss
  2. photogrammetric scan for evaluation of accuracy of implant placement and passivity of final prosthesis
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- partially- guided (PG) implant instalment (Active Comparator): partial guided allow control until the drill before the last one using universal drilling kit and the final osteotomy done with the system specific finishing drill after removal of the surgical guide.
  Interventions: Device: cone beam computed tomography; Device: photogrammetric scan using elite scanner (shining 3d)
- fully- guided (FG)implant instalment (Active Comparator): Fully guided guides allow complete guidance to the drills tell the final one in addition to implants placement through the guide with control to the implant timing
  Interventions: Device: cone beam computed tomography; Device: photogrammetric scan using elite scanner (shining 3d)

INTERVENTIONS:
Device: cone beam computed tomography — -Implant marginal bone height changes will be measured by cone beam radiograph after one and two years of loading
Device: photogrammetric scan using elite scanner (shining 3d) — implant placement accuracy will be evaluated using photogrammetric scan after implant insertion

SUMMARY:
compare fully versus partially guided all on four implants placement immediately loaded by maxillary and mandibular screw retained overdentures: A radiographic and photogrammetric measurement of accuracy of implant position and passivity of superstructures.

The measurements will be done as follows:

1. Photogrammetric scan immediately after implant instalments to measure 3D accuracy of implant position and Passivity of super structure
2. Cone beam X ray to measure the implant marginal bone height changes.
3. Implant marginal soft tissue evaluations including pocket probing depth, plaque and gingival indices. Evaluation will be done immediately, one and two years after loading.

DETAILED DESCRIPTION:
Sixteen healthy, fully edentate patients will be selected from the Prosthodontic Department, Faculty of Dentistry, Mansoura University. The patients will be informing about the protocol of the study and, they will sign a written consent. The study will be ethically approved according to the faculty of dentistry principles.

Sample size and study design A power analysis was made using a computer software (G* power) to detect the prober sample size based on the results of a previous study in which the authors found a significant difference in mesiodistal measurements between two groups (computer guided implant placement Vs conventional implant placement) using a similar study design. The sample size calculation yields a total of 32 implants (16 implants\ each group) using independent samples t-test. The following are details of sample size calculation: effect size= 0.904, Alpha (α)= .050. power (β)= .80

Patient selection i- Completely healed residual alveolar ridges ii- Angle's class I maxillo-mandibular relationship. iii- Sufficient mandibular and maxillary restorative spaces, at least 15mm evaluated by recording a tentative jaw relation.

iv- Adequate bone height in the premaxilla area, and the anterior mandibular area. This will be evaluated radiographically Exclusion criteria included (i) Systemic disorders affecting bone (such as uncontrolled diabetes mellitus and osteoporosis).

(ii) Local or general contraindication for surgical procedures. (iii) History of chemotherapy or radiation therapy to the head and neck area. (iv) Poor neuromuscular co-ordination. (v) TMJ dysfunction and parafunctional habits

1. Construction of conventional complete denture:

   Each patient will receive conventional complete denture and will be delivered and followed to adjust any post operative complains
2. Construction of surgical guide by dual scan technique:

   - According to the virtual 3D planning and surgical guide designing for implant instalment, patients will randomly be divided into two equal treatment groups as follows: Group (I): partially- guided (PG) implant instalment Group (II): fully- guided (FG)implant instalment
3. Photogrammetic scanning:

   For both groups based on the implant planning position and angulation a presurgical 3D printed model with digital analogue spaces will be constructed and scanned using photogrammetric device after connecting the multiunit digital analogues to the printed model in order to be compared to the model formed after implants placement in each group using photogrammetric device.
4. Implant instalments:

   * Flapless surgical protocol will be followed to install the maxillary and mandibular implants for both groups following all on 4 concepts.
   * Post operative medication and home care will be followed for all patients.
5. Construction of screw retained mandibular and maxillary overdentures

   * Scan bodies will be screwed into the implant fixture and will be scanned intraorally
   * The implant superstructure will be virtually planned and will be milled in (or 3D laser printed into cobalt chromium)
   * Artificial teeth will be milled in according to balanced lingualized scheme and mandibular and maxillary screw retained will be fabricated and immediately delivered into the patient mouth within 2-3 days of implant instalment
6. Methods of evaluation:

   * Passivity of superstructure and 3-D accuracy of implant position will be measured immediately after loading by using photogrammetric device.
   * Implant marginal bone height changes will be measured by cone beam radiograph after one and two years of loading
   * Evaluation peri-implant soft tissue changes in form of probing depth, and gingival and plaque indices will be measured immediately, one and two years of implant loading.

ELIGIBILITY:
Inclusion Criteria:

* Completely healed residual alveolar ridges
* Angle's class I maxillo-mandibular relationship.
* Sufficient mandibular and maxillary restorative spaces, at least 15mm evaluated by recording a tentative jaw relation.
* Adequate bone height in the premaxilla area, and the anterior mandibular area. - This will be evaluated radiographically

Exclusion Criteria:

* Systemic disorders affecting bone (such as uncontrolled diabetes mellitus and osteoporosis).
* Local or general contraindication for surgical procedures.
* History of chemotherapy or radiation therapy to the head and neck area.
* Poor neuromuscular co-ordination.
* TMJ dysfunction and parafunctional habits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
accuracy of implant insertion | immediately after implant insertion
  accuracy of implant position will be measured immediately after implant insertion by using photogrammetry scan for implants with multi-unit abutments intra-orally and on the model created from the planned implants and fitting surface of surgical guide, superimposition of both scans will be done using geomagic software to determine deviation in implant positions between both scans (Presurgical and post surgical) for both groups and calculated in fractions of millimeters, the value of deviation found in both semi-guided and fully-guided groups will be compared.

SECONDARY OUTCOMES:
passive fit of final prosthesis | immediately after final restoration insertion
  passivity of final prosthesis will be evaluated by radiography and gap distance will me measured on radiographic software in fractions of millimeters
Marginal bone loss | 24 months after prosthesis insertion
  Implant marginal bone height changes will be measured by cone beam radiograph after one and two years of loading

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shady Mohamed Shady, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Faculty of Dentistry, mansoura, egypt, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: No